CLINICAL TRIAL: NCT05039944
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of SI-B001 as a Single Agent or in Combination With Chemotherapy in the Treatment of Unresectable or Metastatic Digestive System Malignancies (Colorectal and Gastric Cancer)
Brief Title: SI-B001 as a Single Agent or in Combination With Chemotherapy in the Treatment of Digestive System Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company research strategy adjustment
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SI-B001_211
Record Dates: First submitted 2021-08-22; First posted 2021-09-10 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer
Keywords: CRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; IFL protocol; Folfox protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SI-B001_A (Experimental): Patients with unresectable or metastatic gastric cancer, HER2-negative and without standard treatment were treated with SI-B001 monotherapy.SI-B001 is administered by intravenous drip twice weekly (Q2W).
  Interventions: Drug: SI-B001
- SI-B001_B (Experimental): Patients with MSS KRASwt BRAFwt unresectable or metastatic colorectal cancer who had failed conventional chemotherapy combined with EGFR mab were treated with SI-B001 monotherapy.SI-B001 is administered by intravenous drip twice weekly (Q2W).
  Interventions: Drug: SI-B001
- SI-B001_C (Experimental): Patients with MSS KRASwt BRAFwt unresectable or metastatic colorectal cancer who had failed multiple lines of conventional chemotherapy (excluding EGFR monoclonal antibody) were treated with SI-B001 monotherapy.SI-B001 is administered by intravenous drip twice weekly (Q2W).
  Interventions: Drug: SI-B001
- SI-B001 combined with irinetecan_D (Experimental): Patients with MSI-H KRASwt BRAFwt unresectable or metastatic colorectal cancer who had previously failed to receive anti-PD-1 (L1) mab (excluding EGFR mab) in the first or second line were treated with SI-B001 in combination with irinetecan in the third line.SI-B001 is administered by intravenous drip twice weekly (Q2W).
  Interventions: Drug: SI-B001; Drug: Irinotecan
- SI-B001 combined with FOLFIRI or FOLFOX_E (Experimental): Patients with MSI-H KRASwt BRAFwt unresectable or metastatic colorectal cancer who had previously failed first-line anti-PD-1 (L1) mab were treated with SI-B001 in combination with FOLFIRI or FOLFOX for second-line treatment.SI-B001 is administered by intravenous drip twice weekly (Q2W).
  Interventions: Drug: SI-B001; Drug: FOLFIRI Protocol; Drug: FOLFOX Protocol
- SI-B001 combined with irinetecan_F (Experimental): Patients with MSS KRASwt BRAFwt unresectable or metastatic colorectal cancer who had failed standard first-line treatment containing oxaliplatin or irinotecan plus fluorouracil plus or minus bevacizumab were treated with SI-B001 plus irinotecan in the second-line.SI-B001 is administered by intravenous drip twice weekly (Q2W).
  Interventions: Drug: SI-B001; Drug: Irinotecan

INTERVENTIONS:
Drug: SI-B001 — In Arm_A, B and C, the intravenous infusion dose of SI-B001 was single drug RP2D selected in phase I (Q2W); In Cohort_D, E, and F, SI-B001 was divided into two doses, the high dose was the single drug RP2D selected in phase I clinical trial, and the low dose was the second low dose of single drug RP2D, both of which were administered by intravenous infusion.
Drug: Irinotecan — Administration by intravenous infusion, 180 mg/m2 Q2W.
  Arms: SI-B001 combined with irinetecan_D; SI-B001 combined with irinetecan_F
Drug: FOLFIRI Protocol — FOLFIRI is administered intravenously at the standard dose recommended by the guidelines(Q2W).
  Arms: SI-B001 combined with FOLFIRI or FOLFOX_E
Drug: FOLFOX Protocol — FOLFOX is administered intravenously at the standard dose recommended by the guidelines(Q2W).
  Arms: SI-B001 combined with FOLFIRI or FOLFOX_E

SUMMARY:
This multi-center, open label Phase II clinical study is performed in patients with unresectable or metastatic malignant tumors of the digestive system (colorectal cancer, gastric cancer). This study is investigating the safety and efficacy of SI-B001 at monotherapy or optimal combination dose with chemotherapy in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18;
2. Expected survival time ≥3 months;
3. Patients with unresectable or metastatic colorectal cancer or gastric cancer confirmed by histology or pathology:

   Cohort_A: Patients with unresectable or metastatic gastric cancer, HER2-negative, without standard treatment.

   Cohort_B: Patients with MSS KRASwt BRAFwt unresectable or metastatic colorectal cancer, failure of conventional chemotherapy combined with EGFR mab, and withdrawal of EGFR mab for less than 3 months.

   Cohort_C: MSS KRASwt BRAFwt patients with unresectable or metastatic colorectal cancer who have failed multiline conventional chemotherapy (without EGFR monoclonal antibody therapy).

   Cohort_D: MSI-H KRASwt BRAFwt patients with unresectable or metastatic colorectal cancer and previous first - or second-line treatment failure with anti-PD-1 (L1) mab (excluding EGFR mab).

   Cohort_E: MSI-H KRASwt BRAFwt patients with unresectable or metastatic colorectal cancer who have previously failed first-line anti-PD-1 (L1) mab therapy.

   Cohort_F: MSS KRASwt BRAFwt patients with unresectable or metastatic colorectal cancer who have failed standard therapy with first-line oxaliplatin or irinotecan plus fluorouracil plus or minus bevacizumab.
4. No previous anti-EGFR antibody therapy (excluding Cohort_B);
5. Agree to provide 4 specimens (thickness 5μm) of tumor tissue specimens (non-stained sections (anti-removal)) archiving from primary or metastatic tumors;agree to provide 6 unstained sections surgical specimens (anti-removal, thickness 10μm) or fresh tissue samples;
6. There must be at least one measurable lesion conforming to the RECIST V1.1 definition;
7. Cohort_A, B, C fitness scores ≤2, Cohort_D, E, F fitness scores ≤1;
8. Toxicity of previous antitumor therapy has been restored to ≤1 as defined by NCI-CTCAE V5.0 (except for toxicity that the researchers judge to be of no safety risk, such as hair loss, grade 2 peripheral neurotoxicity, and stabilized hypothyroidism after hormone replacement therapy);
9. Organ function levels must meet the following requirements and meet the following standards:

   A) Bone marrow function: absolute value of neutrophil count (ANC) ≥1.5×109/L, platelet count ≥100×109/L (platelet count ≥75×109/L in Patients with Cohort_A, B and C), hemoglobin ≥90 g/L (hemoglobin ≥85 g/L in patients with Cohort_A, B and C); B) Liver function: Total bilirubin TBIL≤1.5×ULN (total bilirubin TBIL≤ 3×ULN in Gilbert's syndrome, liver cancer or liver metastases); AST and ALT ≤2.5×ULN in patients without liver metastasis; AST and ALT ≤5.0×ULN in patients with liver metastasis; C) Renal function: Creatinine (Cr) ≤1.5×ULN, or creatinine clearance (Ccr) ≥50 mL/min (according to Cockcroft and Gault formula); D) Urine routine / 24-hour protein quantification: qualitative urine protein ≤1+ (if qualitative urine protein ≥2+, 24 hours < 1g can be included); E) Cardiac function: left ventricular ejection fraction ≥50%; F) Coagulation function: International standardized ratio (INR) ≤1.5×ULN, and activated partial thrombin time (APTT) ≤1.5×ULN;
10. Eligible patients (male and female) who are fertile must agree to use a reliable contraceptive method (hormonal or barrier method or abstinence, etc.) with their partner during the trial and for at least 6 months after the last medication;Women of childbearing age must have a negative blood or urine pregnancy test within 7 days prior to the first use of the study drug.

Exclusion Criteria:

1. Colorectal cancer patients with HER2 positive (immunohistochemical +++, or immunohistochemical ++ with FISH amplification);
2. Have received chemotherapy, radiotherapy, biotherapy, endocrine therapy, immunotherapy and other anti-tumor therapy within 4 weeks prior to the first use of the study drug, except the following:

   Oral fluorouracil and small molecule targeted drugs are 2 weeks before the first administration of the study drug or within the 5 half-lives of the drug (whichever is longer); The traditional Chinese medicines with anti-tumor indications were within 2 weeks before the first use of the study drug;
3. Received an unmarketed clinical investigational drug or treatment within 4 weeks prior to the first use of the investigational drug;
4. Has undergone major organ surgery (excluding needle biopsy, tracheotomy, gastrostomy, etc.) or has significant trauma within 4 weeks before the first use of study drugs, or needs to undergo elective surgery during the trial;
5. Previous recipients of allogeneic hematopoietic stem cell transplantation or organ transplantation;
6. A history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

   Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, grade iii atrioventricular block, etc.

   In the resting state, QT interval was prolonged (QTc > 450 msec in men or QTc > 470 msec in women); Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other grade 3 or higher cardio-cerebrovascular events within 6 months prior to the first administration; New York Heart Association (NYHA) heart function grade ≥II heart failure;
7. Active autoimmune and inflammatory diseases, such as systemic lupus erythematosus, inflammatory bowel disease, etc., except type I diabetes, hypothyroidism that can be controlled only with replacement therapy, and skin diseases that do not require systemic treatment (e.g., vitiligo, psoriasis);
8. A history of other malignant tumors within 3 years prior to the first administration, with no signs of recurrence and metastasis;
9. Poorly controlled hypertension (systolic blood pressure & GT;150 mmHg or diastolic pressure >100 mmHg);
10. Pulmonary disease defined as grade 3 or higher according to CTCAE V5.0;Patients with past or present interstitial lung disease (ILD);
11. Cerebral parenchymal or meningeal metastases with clinical symptoms are not suitable for inclusion by the investigator;
12. Had ≥ grade 3 infusion-related reactions during prior anti-EGFR antibody therapy (Cohort_B only);
13. There are known allergic contraindications to any excipients of SI-B001 and chemotherapeutic agents selected in this study;
14. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBV-DNA copy number > 104) or hepatitis C virus infection (HCV-RNA > center detection lower limit);
15. Active infections requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.;
16. Pregnant or lactating women;
17. Persons with mental disorders or poor compliance;
18. The investigator considers that the subject has a history of other serious systemic diseases or other reasons and is not suitable to participate in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
ORR | Up to approximately 24 months
  Objective Response Rate
Optimal combination dose (only IIa) | Up to approximately 24 months
  Optimal combination dose of SI-B001 with chemothreapy (only IIa)

SECONDARY OUTCOMES:
PFS | Up to approximately 24 months
  Progression-free Survival
DCR | Up to approximately 24 months
  Disease Control Rate
DOR | Up to approximately 24 months
  Duration of Response
OS | Up to approximately 24 months
  Overall Survival
TEAE | Up to approximately 24 months
  Treatment Emergent Adverse Events
Cmax | Up to approximately 24 months
  Maximum serum concentration
Tmax | Up to approximately 24 months
  Time to maximum serum concentration
Ctrough | Up to approximately 24 months
  Minimum serum concentration
ADA | Up to approximately 24 months
  anti-SI-B001 antibody

CONTACTS AND LOCATIONS:
Overall Officials: Weijian Guo, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China